CLINICAL TRIAL: NCT02605421
Title: Tandem Myeloablative Consolidation Therapy and Autologous Stem Cell Rescue for High-Risk Neuroblastoma
Brief Title: Myeloablative Consolidation Therapy and Tandem Autologous Stem Cell Rescue in Patients With High-Risk Neuroblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015LS108
Record Dates: First submitted 2015-11-12; First posted 2015-11-16 (Estimated); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Neuroblastoma
Keywords: High-risk neuroblastoma; Neuroblastoma; Myeloablative chemotherapy; Myeloablative consolidation chemotherapy; Autologous peripheral blood stem cell rescue; PBSC; Autologous stem cell rescue
MeSH Terms: conditions — Neuroblastoma | interventions — Thiotepa; Cyclophosphamide; Melphalan; Etoposide; Carboplatin; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients Treated for Neuroblastoma (Experimental): Consolidation course #1 consists of thiotepa and cyclophosphamide followed by a PBSC rescue. Consolidation course #2 consists of melphalan, etoposide and carboplatin followed by a second PBSC rescue. Post infusion, patients will receive Granulocyte-Colony Stimulating Factor beginning on Day 0 of each consolidation course.
  Interventions: Drug: Thiotepa; Drug: Cyclophosphamide; Drug: Melphalan; Drug: Etoposide; Drug: Carboplatin; Biological: Autologous Stem Cell Infusion; Biological: Granulocyte colony stimulating factor

INTERVENTIONS:
Drug: Thiotepa — Thiotepa by IV once daily for 3 doses on Days -7, -6 and -5. Given as part of Consolidation Course #1 along with Cyclophosphamide.
Drug: Cyclophosphamide — Cyclophosphamide by IV once daily for 4 doses on Days -5, -4, -3 and -2. Given as part of Consolidation Course #1 along with Thiotepa.
Drug: Melphalan — Melphalan by IV once daily for 3 doses on Days -8, -7, and -6. Given as part of Consolidation Course #2 along with Etoposide and Carboplatin.
Drug: Etoposide — Etoposide by IV once daily for 4 doses on Days -8, -7, -6 and -5. Given as part of Consolidation Course #2 along with Melphalan and Carboplatin.
Drug: Carboplatin — Carboplatin by IV once daily for 4 doses on Days -8, -7, -6 and -5. Given as part of Consolidation Course #2 along with Etoposide and Melphalan.
Biological: Autologous Stem Cell Infusion — On Day 0 the stem cells will be infused immediately after thawing over 15-60 minutes per institutional guidelines.
Biological: Granulocyte colony stimulating factor — Beginning on day 0 after infusion of the PBSC, patients will receive G-CSF SQ or IV (SQ preferred) 5 micrograms/kg once daily and continuing once daily until post-nadir ANC > 2000/μL for 3 consecutive days.
  Other Names: G-CSF

SUMMARY:
This is a phase II single center study to administer two courses of myeloablative consolidation chemotherapy each followed by an autologous peripheral blood stem cell (PBSC) rescue in patients with high-risk neuroblastoma who have completed induction chemotherapy (independent of this study). Ideally, patients should begin consolidation chemotherapy no later than 8 weeks after the start of Induction Cycle #5; however it is strongly recommended to begin consolidation within 4-6 weeks after the start of Induction Cycle #5.

ELIGIBILITY:
* Less than 30 years of age at diagnosis of neuroblastoma
* End of Induction disease evaluation demonstrating CR, PR, MR or SD
* Hematopoietic Recovery from last induction course of chemotherapy
* No uncontrolled infection
* Minimum frozen PBSCs of 2 x 10^6 CD34 cells/kg for each transplant are mandatory and a PBSC of 2 x 10^6 CD34 cells/kg for back-up are strongly recommended (thus, PBSC of no less than 6 x 10^6 CD34 cells/kg is encouraged). These must all be collected prior to the initiation of consolidation.
* Adequate organ function defined as:

  * Hepatic: AST and ALT < 3 x upper limit of institutional normal; ALT ≤ 3 x ULN for age; total bilirubin ≤ 1.5 x ULN for age, if baseline was normal, > 1.0 1.5 x baseline if baseline was abnormal
  * Cardiac: shortening fraction ≥ 27% or ejection fraction ≥ 45%, no clinical congestive heart failure
  * Pulmonary: no evidence of dyspnea at rest and norequirement for supplemental oxygen
  * Renal: Creatinine clearance or GFR > 60 mL/min/1.73m^2. If a creatinine clearance is performed at end induction and the result is < 100 ml/min/1.73m^2, a GFR must then be performed using a nuclear blood sampling method or iothalamate clearance method. Camera method is NOT allowed as measure of GFR prior to or during Consolidation therapy for patients with GFR or creatinine clearance of < 100 ml/min/1.73m^2
* Recovery from acute toxicities of last cycle of induction chemotherapy
* Appropriate written consent - adult or parent/guardian if patient is < 18 years of age and minor information sheet if patient is > 8 years of age

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 3 years from first PBSC infusion
  Percentage of patients with progression free survial. Kaplan-Meier curves and 95% confidence intervals will be used to estimate.

SECONDARY OUTCOMES:
Time to Engraftment | Day 42
  Defined as an absolute neutrophil count (ANC) greater than or equal to 0.5 x 109/L for three consecutive days by day 42 after first transplant.
Relapse | 3 years from first PBSC infusion
  Percentage of patients with relapse. Relapse will be defined as any new lesion; increase of any measurable lesion by >25%; previous negative bone is positive.
Overall Survival | 3 years from first PBSC infusion
  Kaplan-Meier curves and 95% confidence intervals will be used to estimate overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Gupta, MBBS, MPH, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States